CLINICAL TRIAL: NCT01803906
Title: Tissue Study for Mitochondrial Disorders
Brief Title: Tissue Sample Study for Mitochondrial Disorders
Status: Enrolling by invitation | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAAB5754; P01HD032062 (NIH)
Record Dates: First submitted 2012-08-31; First posted 2013-03-04 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Mitochondrial Disorders; Mitochondrial Disease; Melas; Kearns Sayer; NARP; MNGIE; LHON; Mitochondrial Depletion Syndrome; Leigh's Disease
Keywords: mitochondrial disorder; mitochondria; oxidative phosphorylation; oxidative phosphorylation disorders; respiratory chain disorders; mitochondrial disease; melas; kearns sayer; NARP; MNGIE; LHON; Mitochondrial depletion syndrome; Leigh's disease
MeSH Terms: conditions — Mitochondrial Diseases; MELAS Syndrome; Leigh Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any type of tissue could be submitted, however, generally blood, urine, buccal cell (cheek), and muscle are sent.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mitochondrial disease: Patients with known or suspected DNA mutations that affect mitochondrial function. Patients with suspected mitochondrial disorders

SUMMARY:
The investigators are studying patients with undefined mitochondrial diseases to identify genetic mutations in nuclear or mitochondrial Deoxyribonucleic Acid (DNA). Most patients with suspected or known mitochondrial diseases have no genetic confirmation. The investigators expect that evaluating tissue samples from patients with mitochondrial disorders will lead us to discover mutations in new or known genes causing mitochondrial dysfunction.

DETAILED DESCRIPTION:
Presently, the investigators know of about 200 mitochondrial disorders. The investigators know that there are about 1,300 genes responsible for mitochondrial function. Thus, there are a lot of mutated genes to be discovered out there. Currently, most patients with suspected or known mitochondrial disorders do not have genetic confirmation of the disease.

The goal of this project is to perform biochemical and DNA analysis on tissue samples of patients with mitochondrial disorders to find new genes that might be involved in mitochondrial dysfunction.

Leftover patient tissue samples will be obtained for analysis from within the Columbia Presbyterian Medical Center. Left over patient samples may also be sent from outside the institution. This is not a "first-step" in the diagnostic process, but rather an option for evaluation in patient samples for which no known diagnosis or genetic confirmation has been made.

The research laboratory does not guarantee that a sample will be analyzed. Sample analysis is performed according to research interest. If they choose, patients can be contacted should laboratory findings provide insight into their disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of having a mitochondrial disorder
* Patients who may carry a genetic mutation or be related to someone with a genetic mutation which may cause a mitochondrial disorder

Exclusion Criteria:

* Patients who are not suspected of having a mitochondrial disorder

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages, race, gender with known or suspected mitochondrial disorders and their carrier relatives (if requested).
Sampling Method: Non-Probability Sample
Enrollment: 6900 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with reduced respiratory chain enzyme levels | Up to 2 years
  Biochemical studies involving mitochondrial function. The levels will be compared to normal levels.

SECONDARY OUTCOMES:
Number of new genetic mutations | Up to 2 years
  Evaluation of potential genetic interaction in clinical signs and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Michio Hirano, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
When applicable we will submit manuscript (s) describing the findings

REFERENCES:
- See also: Link to general laboratory information — http://www.columbiamitodiagnostics.org